CLINICAL TRIAL: NCT04388579
Title: PRAISE@COVID-19: Screening Patients for a Strategic Shift to Pulmonary Telerehabilitation
Brief Title: Screening Patients for a Strategic Shift to Pulmonary Telerehabilitation Because of COVID-19
Acronym: PRAISE@COVID
Status: Completed | Type: Observational
Sponsor: University of Lisbon (Other)
Collaborators: Centro Hospitalar Lisboa Norte (Other); Fundação para a Ciência e a Tecnologia (Other); Nippon Gases Portugal, Unipessoal, Lda. (Unknown)
Responsible Party: Principal Investigator, Catarina Santos, PhD student, Physiotherapist MSc, University of Lisbon
Other Study IDs: 046i/17
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Disease
Keywords: self-efficacy; PRAISE; Pulmonary Telerehabilitation
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Respiratory Physiotherapy, Exercise Therapy, Patient Education

SUMMARY:
This study applied the Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) on respiratory patients who had their on-going ambulatory Pulmonary Rehabilitation program interrupted due to the COVID-19 outbreak. The research hypothesis is that ranking patients' self-efficacy is a useful screening tool to support patients' follow-up on a Pulmonary Rehabilitation telehealth solution to be explored during the COVID-19 outbreak.

DETAILED DESCRIPTION:
This was an observational study applied to a convenience sample of Pulmonary Rehabilitation outpatients from Hospital Pulido Valente in Lisbon, Portugal, which had ambulatory treatments suspended due to the COVID-19 outbreak. Cross-sectional design was operationalized by a physiotherapist who promptly screened by phone a sample of 100 patients, assessing 90% of the eligible population. Patients had no previous therapeutic relation with the physiotherapist, who was also blind to patient's status at the Pulmonary Rehabilitation program. The screening call took a mean time of 484.8 ± 173.6 seconds, which is proximately about 8 ± 3 minutes per patient, with a minimum of 5 and a maximum of 19 minutes. Screening process included applying the Portuguese version of the Pulmonary Rehabilitation Adapted-Index of Self-Efficacy (PRAISE) and also included questioning patients if they were engaging on a daily routine of respiratory exercises by their initiative, and also if they managed to preserve a daily period to practice physical activity. In case of a positive answer, information concerning available equipment and exercise protocol adopted at patient's home environment was also collected. On a subsequent phase, data about patients' age, diagnosis referral for Pulmonary Rehabilitation, number of completed treatment sessions and weekly frequency, was collected from the hospital information system. Statistical analysis and data management were performed using the Statistical Package for the Social Sciences (SPSS) version 25.0 (SPSS Inc., Chicago, IL, USA). A formal sample size was not calculated since this was a convenience sample of 100 patients. Descriptive statistics included mean, standard-deviation, median, quartiles, range, minimum and maximum values and frequencies presented as percentages. Inferential statistics included the Pearson coefficient for PRAISE, age and number of treatment sessions, with the remaining variables analysed by the Spearman coefficient. PRAISE was the primary outcome, with mean comparison analysed by the Student t test, proved the normal distribution and equal variances. A p value of less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute respiratory disease
* Patients with chronic respiratory disease
* Patients attending a hospital-based Pulmonary Rehabilitation program

Exclusion Criteria:

* Cognitive deficit for answering a questionnaire

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adults attending an outpatient Pulmonary Rehabilitation program based at Hospital Pulido Valente from Centro Hospitalar Universitário Lisboa Norte, in Lisbon, Portugal
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Patient's self-efficacy | 3 days
  Vincent and co-authors (2011) proposed the Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE). The PRAISE tool is composed by a total of 15 items, combining 10 items from the General Self-Efficacy Scale (GSE) by Schwarzer and Jerusalem (1995), and 5 new specific items related to Pulmonary Rehabilitation. Each item is scored from 1 to 4 with a total range from 15 to 60, with higher scores indicating higher levels of self-efficacy. This study applies the Portuguese PRAISE version by Santos CD and co-authors (2019).

SECONDARY OUTCOMES:
Respiratory exercises | 3 days
  Patients were questioned if they were engaging on a daily routine of respiratory exercises by their initiative while isolated at home COVID-19 outbreak. The answer was registered as yes/no.
Physical activity | 3 days
  Patients were questioned if they managed to preserve a daily period to practice physical activity while isolated at home during COVID-19 outbreak. The answer was recorded as yes/no. In case of a positive answer, information concerning available equipment and exercise protocol adopted at patient's home environment was also collected.

OTHER OUTCOMES:
Treatment sessions completed | 3 days
  Number of Pulmonary Rehabilitation hospital sessions completed as outpatient, according to Hospital Pulido Valente information system
Treatment weekly frequency | 3 days
  Number of Pulmonary Rehabilitation sessions planned per week, according to Hospital Pulido Valente information system

CONTACTS AND LOCATIONS:
Overall Officials: Catarina D Santos, MSc, Principal Investigator — University of Lisbon; Cristina Bárbara, PhD, Study Director — University of Lisbon
Locations (3):
- Portugal (3):
  - Nippon Gases Portugal Unipessoal Lda, Maia, Porto District
  - Universidade de Lisboa, Faculdade de Medicina, Instituto de Saúde Ambiental (ISAMB), Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, Hospital Pulido Valente, Unidade de Reabilitação Respiratória, Lisbon

IPD SHARING:
Plan to Share IPD: No